CLINICAL TRIAL: NCT03307889
Title: SOMNOmedics Clinical Validation Trial of Pulse Transit Time (PTT) Compared With Arterial Line in Patients Undergoing Nonvascular Surgery.
Brief Title: SOMNOmedics Clinical Validation Trial
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Michael Hultström, Associate professor, Uppsala University
Other Study IDs: EPN dnr 2017/068
Record Dates: First submitted 2017-10-06; First posted 2017-10-12 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Blood Pressure; Perioperative/Postoperative Complications
Keywords: perioperative monitoring
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Observational study in which pulse transit time (PTT) as a method and the device to register this data is compared with arterial blood pressure.

The population is composed of pediatric and adult patients in anesthesia or intensive care in need of arterial blood pressure monitoring.

DETAILED DESCRIPTION:
Plan to enroll patients who accept the terms of the study consecutively. The population is composed by pediatric and adult patients in anesthesia and intensive care in need of close blood pressure monitoring.

After informed consent from the patients themselves, patient and parents and sometimes only parents.

The device measuring PTT is the prepared and calibrated with existing arterial blood pressure. Data is then recorded via the storage capacity of the device and via videocamera. The videocamera is used to identify large disturbances in data registration. This is to identify confounding data and in the end calibrate the device to be more accurate.

Data from the PTT device and the camera is then downloaded to the study computer and to an external hard drive in order to create redundancy in data storage.

Data is then analysed to compare the difference between data recorded from the PTT device and arterial pressure respectively. Aim is to be able to collect sufficient data to be able to decide wether to recommend or advice against clinical use.

Patient data is registered and then handled by our departmental clerk. Data is stored for ten years.

ELIGIBILITY:
Inclusion Criteria:

* Arterial line planned or existing

Exclusion Criteria:

* suspected major perioperative hemodynamic variation.
* non existing consent.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric and adult patients in anesthesia or intensive care.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-08-20 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of pulse transit time (PTT) estimation of blood pressure against intra arterial measurement. | 45 minutes- 120 minutes
  Difference in mmHg between blood pressure calculated by PTT and arterial blood pressure. A video will record the measurement session in order to determine any action correlating to changes in blood pressure. A second use of the video is to determine what other action taken around the patient causing noise or confounding measurements,

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hultström, Ass Prof, Principal Investigator — Uppsala University
Locations (1):
- Akademiska Sjukhuset, Uppsala, Upp, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Anonymous data will be made available to interested researchers after publication. The patients are informed of this fact.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Supporting information will be made available after publication.
Access Criteria: Data and supporting information will be made available to interested researchers upon request.